CLINICAL TRIAL: NCT04654338
Title: Electively Combining Two Ablative RadioTherapy Treatments for Favorable Risk Prostate Cancer Patients (EARTH)
Brief Title: 2 Ablative RadioTherapy Treatments for Prostate Cancer
Acronym: EARTH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Andrew Loblaw, GU Radiation Oncology Site Group Lead, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3592
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Radiation: SABR + HDR

INTERVENTIONS:
Radiation: SABR + HDR — One SABR treatment + one HDR brachytherapy treatment

SUMMARY:
Favorable-risk prostate cancer represent a large proportion of patients diagnosed with prostate cancer and image guided radiation therapy (IGRT) is commonly used to treat these patients using protracted courses of up to 39 treatments over 8 weeks. Stereotactic ablative body radiotherapy (SABR) protocols hold the promise of more convenience, less side effects, less cost and improved system capacity without sacrificing excellent cancer control rates. By the same token, prostate high-dose rate (HDR) brachytherapy boost has been shown to be superior to standard external beam radiation. While two HDR fractions appear to optimize patient convenience and outcomes while minimizing costs, we wanted to determine the tolerability of combining one MR-guided HDR treatment with one SABR treatment to further reduce HDR resource use while maintaining favourable treatment outcomes.

DETAILED DESCRIPTION:
Pre-Treatment:

Planning CT and mpMRI imaging for SABR TRUS with biopsy and insertion of Gold Seed Fiducial Markers Biobanking of urine, blood and biopsy tissue (as per REB#079-2006 Odette Cancer Centre (OCC) biobanking protocol)

Stereotactic Ablative Body Radiation (SABR):

13.5Gy x 1 to whole prostate + 1cm seminal vesicles 2 weeks post-planning, treatment will be delivered as per standard treatment protocols on SABR-compatible linear accelerator with a six-degree of freedom couch. Cone-beam CT imaging will be performed using the implanted fiducials to set up each treatment. All dosimetric parameters will be recorded.

Inter-treatment (approx 1 week post-SABR):

Planning mpMRI and TRUS imaging for HDR Biobanking of urine and blood (as per REB#079-2006 OCC biobanking protocol)

HDR brachytherapy:

13.5 Gy x 1 to the prostate, <20 Gy to DIL Approx 2-3 weeks post-SABR, the HDR dose prescription of 13.5 Gy to the whole gland and <20 Gy to MRI visible lesion will be delivered in one fraction, assuming that dose constraints to critical organs can be met. All dosimetric parameters will be recorded

Patient Assessments / Follow-up Time zero will be the date of SABR treatment. Baseline rectal, urinary and sexual function will be recorded prior to treatment. Acute toxicities will be assessed at 6, 12 and 24 weeks and late toxicities will be assessed at month 9, 24 and every 6 months until year 5 using the Common Terminology Criteria Adverse Events, V 4.0. Bloodwork (PSA and testosterone) and International Prostate Symptom Score (IPSS) evaluations will be performed at baseline week 6, month 3, 6, 9 and 24, and every 6 months until year 5. QOL using the Expanded Prostate Cancer Index Composite (EPIC), EQ-5D and PORPUS questionnaires will be obtained at baseline, month 3, 6, 9 and 24 and every 6 months until year 5. Post-treatment biobanking will be done at 13 and 52 weeks (as per REB#079-2006 OCC biobanking protocol)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Favorable risk disease defined as either:

  * Low risk disease: T1-T2c, grade group 1, PSA < 10 ng/ml or
  * Favorable intermediate risk disease: One of T2c, grade group 2, or PSA 10-20 ng/ml. Patients cannot have percent core positivity > 50%
* Prostate volume < 60 cc as determined by US, CT or MRI
* Ability to undergo MR imaging
* Provide written informed consent

Exclusion Criteria:

* Documented nodal or distant metastases
* Previous pelvic radiotherapy
* Previous transurethral resection of prostate, previous prostatectomy or HIFU
* Use of androgen deprivation therapy. Use of 5-alpha-reductase inhibitors permitted
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >15
* Contra-indication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
* Significant medical co-morbidity rendering patient unsuitable for general anaesthesia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2028-07-29 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicities | 6 months
  Acute GU and GI toxicities according to the NCI CTCAE v4.0

SECONDARY OUTCOMES:
Late Toxicities | 5 years
  Late GU and GI toxicities according to the NCI CTCAE v4.0
QOL | 5 years
  Quality of life changes utilizing the Expanded Prostate Index Composite (EPIC)
PSA | 5 years
  Biochemical failure and PSA kinetics using PSA response rate

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No